CLINICAL TRIAL: NCT06458244
Title: The Efficacy of Allogeneic Hematopoietic Stem Cell Transplantation in Newly Diagnosed High-relapse-risk Core-binding-factor Acute Myeloid Leukemia
Brief Title: The Efficacy of Allo-HSCT in ND HR-CBF-AML
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Shen yang, Chief physician, Ruijin Hospital
Other Study IDs: CBF-AML01
Record Dates: First submitted 2024-01-09; First posted 2024-06-13 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: core binding factor; high-risk; newly diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Drug Therapy; Cytarabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples including bone marrow cells, blood or DNA/RNA extracted from the cells will be reposited for 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- HSCT-group: The participants receive HSCT after two-cycle of consolidation treatment.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation
- Chemo-group: The participants receive chemotherapy after two-cycle of consolidation treatment.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Allogeneic Hematopoietic Stem Cell Transplantation
  Groups: HSCT-group
Drug: Chemotherapy — Chemotherapy for AML consolidation treatment
  Other Names: High-dose cytarabine
  Groups: Chemo-group

SUMMARY:
For newly diagnosed high-relapse-risk core-binding-factor acute myeloid leukemia participants, the investigators aim to perform allogeneic hematopoietic stem cell transplantation after participants finished one cycle of induction and two cycles of consolidation. To access whether the therapeutic regimen is effective for high-relapse-risk core-binding-factor acute myeloid leukemia, the disease-free-survival (DFS), overall survival (OS), non-relapse-mortality of participants is evaluated.

DETAILED DESCRIPTION:
High-relapse-risk definition:

Participants with high-risk gene mutations or complex karyotypes for disease recurrence, or flow cytometry/gene MRD positivity after two chemotherapy treatments; High-risk gene mutations include: TP53, RTK/RAS signaling (FLT3, NRAS, KRAS, KIT, JAK2, CSF3R), chromatin modification (ASXL1, ASXL2, KMD6A, EZH2, SETD2) or mutations listed as intermediate-risk or high-risk in the 2022NCCN guidelines; The positive threshold for flow cytometry MRD was 0.0001%; The MRD threshold of molecular biology is the lowest value of the detection protocol of the center.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with confirmed CBF-AML. Diagnostic criteria include the presence of t(8; 21)(q22; q22)/RUNX1-RUNX1T1 fusion gene detected at the molecular level; or chromosome presence of inv(16)(p13.1q22)/t(16; 16)(p13.1; q22) /Detection of CBFβ-MYH11 fusion gene at the molecular level;
2. Participants with high-risk gene mutations or complex karyotypes for disease recurrence, or flow cytometry/gene MRD positivity after two chemotherapy treatments; High-risk gene mutations include: TP53, RTK/RAS signaling (FLT3, NRAS, KRAS, KIT, JAK2, CSF3R), chromatin modification (ASXL1, ASXL2, KMD6A, EZH2, SETD2) or mutations listed as intermediate-risk or high-risk in the 2022NCCN guidelines; The positive threshold for flow cytometry MRD was 0.0001%; The MRD threshold of molecular biology is the lowest value of the detection protocol of the center.
3. Medical history and diagnosis of MICM, exclusion of MDS, transformation and treatment-related AML;
4. Age 18-65 years old (18 years old ≤Age< 65 years old);
5. Liver and kidney function: blood bilirubin ≤ 35 μmol/L, AST/ALT below 2 times the upper limit of normal, serum creatinine ≤ 150 μmol/L;
6. Normal cardiac function (EF≥50%, New York Cardiac Function Classification NYHA I/II);
7. Physical condition score 0-2 (ECOG score);
8. For participants with peripheral blood leukocytes < 50*109/L at the initial onset, no chemotherapy has been given except for hydroxyurea before the start of induction therapy;
9. For participants with peripheral blood leukocytes ≥ 50*109/L at the initial onset, cytarabine and hydroxyurea are allowed to be treated before the start of induction therapy;
10. Non-pregnant and lactating women;
11. For all women of childbearing age, a pregnancy test must be performed to measure hCG to rule out pregnancy;
12. Obtain informed consent signed by the patient or family member.

Exclusion Criteria:

1. MDS-converted AML, treatment-related AML; mixed cell leukemia; AML with central nervous system infiltrates and extramedullary lesions at the time of onset;
2. Relapse AML;
3. Allergies or contraindications to any of the drugs involved in the protocol;
4. Liver and kidney function are obviously abnormal, exceeding the enrollment criteria;
5. Cardiac disease: including echocardiogram EF <50%, cardiac insufficiency (New York cardiac function classification NYHA: III/IV), pericardial effusion (CTCAE score >2) within six months after acute myocardial infarction, ECG QTc >470ms;
6. Lung diseases: pulmonary edema, pleural effusion (CTCAE score >2);
7. Suffering from malignant tumors of other organs at the same time;
8. Active patients with HAV, HBV, HCV and tuberculosis, HIV-positive patients;
9. Concomitant other hematologic diseases (including coagulation abnormalities unrelated to leukemia);
10. Inability to understand or follow the study protocol;
11. Those who participate in other clinical studies at the same time; Presence of any other condition that would preclude the conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly Diagnosed High-relapse-risk Core-binding-factor Acute Myeloid Leukemia in Ruijin Hospital
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
disease-free-survival | from data of AML diagnosis until the data of AML relapse, assessed up to 3 years
  disease-free-survival
The relation of CBF-AML genetics subgroup with MRD negativity rate after chemotherapy and DFS after transplantation | from data of AML diagnosis until the data of CR-achieved status, assessed up to 3 years
  The relation of CBF-AML genetics subgroup with MRD negativity rate after chemotherapy and DFS after transplantation

SECONDARY OUTCOMES:
Rate of non-relapse-mortality | the data of death from any cause, assessed up to 3 years
  the ratio of non-relapse-mortality cases and all the mortality cases
overall survival | from data of AML diagnosed until the data of death from any cause, assessed up to 3 years
  overall survival
adverse events | from enrollment to study completion, a maximum of 3 years
  adverse events related with the indicated regimen

CONTACTS AND LOCATIONS:
Overall Officials: Yang Shen, MD, PhD, Study Director — Ruijin Hospital, Shanghai, China
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No